CLINICAL TRIAL: NCT01849536
Title: Corneal Biomechanics and Continuous IOP Monitoring Using Soft Contact Lenses in Glaucomatous Patients
Acronym: BIOLENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2012/20
Record Dates: First submitted 2013-04-26; First posted 2013-05-08 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Open Angle Glaucoma With a Progressive Visual Field
Keywords: Open angle glaucoma; Corneal biomechanics; Intra ocular pressure; IOP; IOP fluctuation; Continuous IOP monitoring; SENSIMED Triggerfish®
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SENSIMED Triggerfish® (Experimental): SENSIMED Triggerfish®
  Interventions: Device: SENSIMED Triggerfish®

INTERVENTIONS:
Device: SENSIMED Triggerfish®

SUMMARY:
Ocular hypertension and its fluctuations is a major risk factor of glaucoma onset and progression. In normal eyes, IOP presents a circadian rhythm, but in glaucomatous eyes IOP circadian rhythm is altered and varied widely between patients. To date, the only way to evaluate 24 hour IOP fluctuations is a regular GAT-IOP measurement during a 24-hour hospitalization. This method is expensive and does not reflect physiological conditions because it requires IOP measurements during sleeping periods that may potentially produce artifacts.

Sensimed AG has developed a new medical device SENSIMED Triggerfish® that enables a 24-hour continuous monitoring of IOP fluctuations. As any IOP measurements methods, this medical device might be influenced by corneal properties of the cornea as central corneal thickness, keratometry or biomechanics. We, therefore, investigate the corneal lens tolerance, potential modifications of corneal parameters after a 24-hour wear of the lens, and its influence on data collected during the whole period of analysis. Then we will also analyze the influence of corneal parameters on continuous IOP fluctuations measured with the contact sensor and finally the correlation between data collected and the rate of progression (severity) of glaucoma evaluated with visual field test or optic nerve head damages.

ELIGIBILITY:
Inclusion Criteria:

* At least 40 year-old
* Signed informed consent
* Visual field defect : at least 2 visual field already done, only the second one is considered for the visual field defect diagnosis, using theses criterion:

  * 3 adjacent points with at least 5db loss
  * Or 1 point with at least 10 db loss
  * Or a 10db difference between two adjacent points on either sides of the nasal horizontal meridian
* Open angle glaucoma patients with a progressive visual field
* For women of childbearing potential, adequate contraception

Exclusion Criteria:

* Corneal dystrophy, scars or corneal surgery
* Iridocorneal angle opening less than 3 using Shaeffer classification
* History of glaucoma surgery
* Any contraindications with the SENSIMED Triggerfish® device, as written in the user manual (active eye disease, severe dry eye, contraindications for silicone contact lens wear…)
* Diabetes
* Sleep Apnea Syndromes
* Cataract surgery
* High myopia
* Pregnancy and lactation
* Patients not able to understand the character and individual consequences of the investigation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Corneal biomechanics influence on IOP fluctuation. | 24h
  To evaluate corneal biomechanics influence on IOP fluctuation using SENSIMED Triggerfish® for glaucoma patients with a progressive visual field.

SECONDARY OUTCOMES:
Correlation between visual field defects and IOP fluctuations measurements. | 24h
  To evaluate the correlation between visual field defects and IOP fluctuations measurements.
Correlation between the severity of optic nerve head damages and IOP. fluctuations measurements | 24h
  To evaluate the correlation between the severity of optic nerve head damages measured with OCT and IOP fluctuations measurements.
Lens tolerance and corneal parameters after 24-hours of contact lens wear. | 24h
  To evaluate lens tolerance and corneal parameters after 24-hours of contact lens wear (Pachymetry, Corneal hysteresis and Keratometry ).

CONTACTS AND LOCATIONS:
Overall Officials: Cédric SCHWEITZER, MD, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Service d'ophtalmologie Hôpital Pellegrin, CHU de Bordeaux, Bordeaux, France